CLINICAL TRIAL: NCT00151931
Title: A Multi-Centre, Open-Label Study Assessing the Efficacy and Tolerability of Lanthanum Carbonate in the Reduction of Serum Phosphate Levels in End Stage Renal Disease Patients Receiving Dialysis
Brief Title: Efficacy and Tolerability of Treatment With Lanthanum Carbonate in Patients With End Stage Renal Disease Receiving Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD405-313
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — lanthanum carbonate

INTERVENTIONS:
Drug: Lanthanum carbonate

SUMMARY:
The purpose of this study is to assess phosphate reduction and control in patients with End Stage Renal Disease treated with lanthanum carbonate

ELIGIBILITY:
Inclusion Criteria:

* Males and females of childbearing potential agree to take adequate precautions to prevent contraception
* Patients diagnosed with ESRD must have been receiving a stable dialysis regimen for chronic renal failure for the 2 consecutive months prior to enrollment in the study
* Patient requires treatment for hyperphosphataemia

Exclusion Criteria:

* Pregnant or lactating women
* Patients who continue to require treatment with compounds containing calcium, aluminum or magnesium
* Patients with clinically significant uncontrolled concurrent illness, a life-threatening malignancy or current multiple myeloma
* Patients who are HIV+
* Patients with any significant gastrointestinal surgery or disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456
Dates: Start 2004-05-11 (Actual); Primary Completion 2006-01-12 (Actual); Study Completion 2006-01-12 (Actual)

PRIMARY OUTCOMES:
Change in pre-dialysis serum phosphate levels at Week 3 compared with Week 5 | Week 3 and Week 5

SECONDARY OUTCOMES:
Treatment emergent adverse events | Throughout the study period of approximately 20 months.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

REFERENCES:
- [Background] Hutchison AJ, Laville M; SPD405-313 Lanthanum Study Group. Switching to lanthanum carbonate monotherapy provides effective phosphate control with a low tablet burden. Nephrol Dial Transplant. 2008 Nov;23(11):3677-84. doi: 10.1093/ndt/gfn310. Epub 2008 Jun 24. PMID 18577536
- See also: FDA Recall Information — http://www.fda.gov/opacom/7alerts.html